CLINICAL TRIAL: NCT00004811
Title: Phase I/II Study of Itraconazole for Blastomycosis, Histoplasmosis, and Sporotrichosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Alabama at Birmingham (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12013; NIAID-MSG-6A
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2001-12

CONDITIONS: Histoplasmosis; Sporotrichosis; Blastomycosis
Keywords: blastomycosis; fungal infection; histoplasmosis; immunologic disorders and infectious disorders; rare disease; sporotrichosis
MeSH Terms: conditions — Histoplasmosis; Sporotrichosis; Blastomycosis; Mycoses; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Itraconazole

INTERVENTIONS:
Drug: itraconazole

SUMMARY:
OBJECTIVES: I. Evaluate the tolerance of patients with blastomycosis, histoplasmosis, and sporotrichosis to different doses of itraconazole (R51,211).

II. Determine levels of itraconazole in serum and other body fluids. III. Assess the course of illness during itraconazole therapy. IV. Determine the dosage of itraconazole that is safe and well tolerated by 80%-90% of patients and estimate the potential of this dosage for use in future comparative trials.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a study to estimate the optimal dose of oral itraconazole. Patients are treated at 1 of 3 doses of itraconazole; the starting dose for each patient is determined at entry.

Therapy is administered daily for 3-6 months. Patients with progressive disease may be treated at the next higher dose; there may be only 1 such increase. Concurrent systemic and topical antifungals are prohibited.

Patients are followed at 1, 3, 6, and 12 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Culture-proven fungal disease, i.e.: Chronic cavitary histoplasmosis Extrapulmonary histoplasmosis, e.g., mucosal disease Blastomycosis Sporotrichosis Positive culture after last dose of any prior therapy Requires antifungal therapy with amphotericin B or ketoconazole No fungal meningitis No central nervous system disease No immediately life-threatening disease --Prior/Concurrent Therapy-- At least 1 month since therapy for same disease No more than 2 mg/kg prior amphotericin B (total dose) No more than 2 mg/kg prior ketoconazole (total dose) No concurrent immunosuppressives, including: Corticosteroids Azathioprine Cytotoxic agents --Patient Characteristics-- Hepatic: AST no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Bilirubin no greater than 3 mg/dL Other: No acquired immunodeficiency syndrome No pregnant or nursing women Effective contraception required of fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7
Dates: Start 1985-03

CONTACTS AND LOCATIONS:
Overall Officials: William Dismukes, Study Chair — University of Alabama at Birmingham